CLINICAL TRIAL: NCT05206422
Title: DORAYA-HF: Assessment of the Doraya Catheter for the Treatment of Volume Overload in Acute Heart Failure Patients With Insufficient Response to Diuretics
Brief Title: DORAYA-HF Early Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Revamp Medical Inc. (Industry)
Responsible Party: Sponsor
Organization: Revamp Medical Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIS-D-03
Record Dates: First submitted 2021-12-28; First posted 2022-01-25 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Acute Decompensated Heart Failure
Keywords: ADHF

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Control Arm (No Intervention): Diuretics only
- Doraya Catheter (Experimental): Doraya Catheter with diuretics
  Interventions: Device: Doraya Catheter

INTERVENTIONS:
Device: Doraya Catheter — The Doraya Catheter is a temporary intravenous flow regulator, positioned in the inferior vena cava below the level of the renal veins
  Arms: Doraya Catheter

SUMMARY:
The study objective is to evaluate the feasibility of the Doraya Catheter and measure clinical performance and safety endpoints, in ADHF patients deemed to have insufficient diuretic response.

ELIGIBILITY:
INCLUSION.

1. Subject is >18 years of age.
2. Subject is hospitalized with primary diagnosis of ADHF.
3. N-terminal-pro-brain natriuretic peptide (NT-proBNP) ≥1,000 pg/m or BNP≥250 pg/mL for body-mass index (BMI) ≤25.
4. Evidence of fluid overload as indicated by 2 or more of the following criteria:

   1. peripheral edema ≥ 2+
   2. radiographic pulmonary edema or pleural effusion
   3. enlarged liver or ascites
   4. pulmonary rales or paroxysmal nocturnal dyspnea, or orthopnea
   5. Jugular venous distention > 7 cmH2O
5. IVCCI < 50% by cardiac ultrasonography or elevated CVP (or RAP) ≥12 mmHg (Invasively measured).
6. Subject insufficiently responds to IV diuretic therapy defined as average hourly urine output <125ml/hour over 6 hours OR cumulative urine output < 3L over 24 hours OR a Net Fluid Loss <375mL in a 12-hour timeframe following ≥2 diuretic challenges with a minimum of:

   1. 1st diuretic dose: ≥2X chronic oral daily dose (IV) or 80 mg IV Lasix or equivalent.
   2. 2nd diuretic dose: ≥ 80 mg IV Lasix or equivalent.
7. Females who are not pregnant or lactating and not planning to become pregnant for the duration of the study. Females of child-bearing potential must have a negative pregnancy test.

   Procedural Inclusion Criterion
8. CVP (or RAP) ≥12 mmHg and PCWP ≥ 18 mmHg confirmed in the Cath Lab, via femoral line, pigtail, Swan Ganz, or other indwelling catheter.

EXCLUSION

1. Systolic blood pressure <90 mmHg at the time of screening.
2. Acute myocardial infarction or acute coronary syndrome or cardiogenic shock or pleurocentesis within past 14 days or cardiovascular intervention within past 14 days.
3. Known LVEF < 10% by echocardiography within 1 year prior to enrollment.
4. Complex congenital heart disease (e.g., Tetralogy of Fallot subjects, single ventricle physiology).
5. Known active myocarditis, hypertrophic obstructive cardiomyopathy, infiltrative cardiomyopathy (e.g., amyloidosis), constrictive pericarditis or cardiac tamponade.
6. Severe Aortic valvular disorder (i.e., hemodynamically relevant valvular diseases such as severe stenosis \severe regurgitation) or Severe mitral disease with planned intervention.
7. Subject has severe renal dysfunction, defined as either eGFR <25 ml/min/1.73 m2 BSA on admission or on renal replacement therapy.
8. Subject with advanced liver disease: either Total Bilirubin > 4 mg/dL or Serum sodium (corrected for glucose) < 125 mmol/L.
9. Treatment with high dose IV inotropes within 2 days prior to enrollment. High dose is defined as > 1 unit of inotrope (excluding Digoxin) as follows: 5 µg/kg/min dopamine = 1 unit, 5 µg/kg/min dobutamine= 1 unit, 0.375 µg/kg/min milrinone = 1 unit.
10. Subject with a history of:

    1. Deep vein thrombosis that occurred < 6 months prior to enrollment, and/or;
    2. Pulmonary embolism episode that occurred < 6 months prior to enrollment.
11. Evidence of active systemic infection documented by either one of the following: fever >38°C/100°F, or ongoing uncontrolled infection (i.e. inflammatory parameters not decreasing despite > 48 hrs of antibiotic treatment).
12. Subjects with a known infra-renal IVC diameter of <16mm.
13. Moribund subject or subject with severe or deteriorating damage in more than 3 critical body systems, based on investigator's clinical judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events | 30 days
  Device or procedure related SAEs rate (including MACE) based on CEC adjudication.
Urine Output | baseline [pre intervention] and accumulated through 24 hours [T=0-24 hours]
  Change in rate of urine output

CONTACTS AND LOCATIONS:
Overall Officials: Mike Favet, Study Director — CEO
Locations (16):
- United States (16):
  - Zuckerberg San Francisco General, San Francisco, California
  - San Francisco VA, San Francisco, California
  - UCSF, San Francisco, California
  - Cleveland Clinic, Weston, Florida
  - Piedmont Hospital, Augusta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Henry Ford, Detroit, Michigan
  - Christian Hospital, St Louis, Missouri
  - UMC of Southern Nevada, Las Vegas, Nevada
  - The Christ Hospital, Cincinnati, Ohio
  - The MetroHealth System, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Oklahoma Heart, Oklahoma City, Oklahoma
  - Prisma Health, Columbia, South Carolina
  - Baylor University Medical Center, Dallas, Texas
  - CHI St. Luke's Health-Baylor St. Luke's Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided